CLINICAL TRIAL: NCT00598338
Title: A Two-Period, Double-Blind, Placebo-Controlled Trial to Evaluate the Effects of re-Treatment of Prucalopride on Efficacy and Safety in Subjects With Chronic Constipation.
Brief Title: Efficacy and Safety Study of Prucalopride for the Re-Treatment of Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-USA-28
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 1
Other: Placebo — o.d.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in the re-treatment of chronic constipation.

Hypothesis:

Retreatment is as effective and safe as treatment with prucalopride in patients with chronic constipation.

DETAILED DESCRIPTION:
This is a multicentre, Phase III trial with a parallel-group design, consisting of a 2 week drug-free run-in period, followed by a 4-week double-blind, placebo-controlled treatment period, a drug-free washout period of at least 2 weeks, and a second 4-week double-blind treatment period.

During the initial run-in period, the subject's bowel habit will be documented in a daily diary and the existence of constipation will be confirmed. Eligible subjects will be randomly allocated to double-blind treatment with either 4 mg prucalopride or placebo, given orally once daily before breakfast, for 4 weeks.

After 4 weeks of treatment, each subject will enter a drug-free washout period. The length of the washout period will be either 2 or 4 weeks, depending on how long it takes for the subject to meet the criteria for constipation. If the subject is unable to re-qualify after a 4-week washout, the subject must be discontinued from the trial.

Subjects who qualify for the second double-blind treatment period will receive the same treatment as during the first treatment period, once-daily for an additional four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant, non-breast-feeding female outpatients at least 18 years of age (no upper age limit).
2. History of constipation; the patient reported having, on average, 2 or fewer spontaneous bowel movements per week that resulted in a feeling of complete evacuation as well as the occurrence of one or more of the following for at least 6 months before the selection visit:

   * very hard (little balls) and/or hard stools at least a quarter of the stools;
   * sensation of incomplete evacuation following at least a quarter of the stools;
   * straining at defecation at least a quarter of the time. The above criteria were only applicable for spontaneous bowel movements, i.e. not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.

   Patients who never had spontaneous bowel movements were considered to be constipated and were eligible for the study.
3. Having functional constipation. Constipation that was not induced by secondary causes of constipation (see exclusion criteria 1 through 7).
4. Willing and able to fill out his/her own diary and questionnaires without help, and able to read and write English.
5. Written informed consent, signed by the patient or legally acceptable representative and by the investigator.
6. Availability for follow-up during the study period as determined in the protocol.

Exclusion Criteria:

1. Patients in whom constipation was thought to be drug-induced, or who were using any disallowed medication
2. Patients with insulin-dependent diabetes mellitus.
3. Patients suffering from endocrine disorders.
4. Patients suffering from neurologic disorders
5. Presence of a megacolon/megarectum or a diagnosis of pseudo-obstruction.
6. Constipation as a result of surgery.
7. Known or suspected organic disorders of the large bowel (i.e. obstruction, carcinoma, or inflammatory bowel disease). Results of a barium enema with flexible sigmoidoscopy or of a colonoscopic examination performed within the last 12 months were needed to rule out organic disorders. A colonoscopic examination or barium enema with flexible sigmoidoscopy performed within the last 3 years was acceptable if the examination was performed for an evaluation of constipation, and there was no history or evidence of weight loss, anaemia, or rectal bleeding, and the patient had 3 consecutively negative stool occult blood tests at screening. Patients with polyps discovered by colonoscopy that were untreated (i.e. by polypectomy) were to be excluded.
8. Presence of known serious, uncontrolled illnesses: clinically significant cardiac, vascular, pulmonary, endocrine, psychiatric disorders (including active alcohol or drug abuse) or metabolic disturbances.
9. Clinically significant cancer within the past 5 years.
10. Subjects known to be HIV positive.
11. Impaired renal function, i.e. serum creatinine concentration >2 mg/dL (>180 micromol/L) or creatinine clearance ≤50 mL/min.
12. Clinically significant abnormalities of haematology, urinalysis, or blood chemistry.
13. Females of child-bearing potential without adequate contraceptive protection during the study. Oral contraceptives, Depo Provera® and Norplant® had to be used for at least 3 months prior to randomisation. Intrauterine devices (IUDs), sterilization, or a double barrier method were other acceptable methods of birth control.
14. Treatment with an investigational drug in the 30 days preceding the run-in phase of the study.
15. Previous treatment with either prucalopride formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 1999-04; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of subjects with three or more spontaneous, complete bowel movements per week. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miner, Jr. B Miner, MD, Principal Investigator — Oklahoma Foundation for Digestive Research